CLINICAL TRIAL: NCT01735383
Title: An Open Label, Balanced, Randomized, Single-dose, Two-treatment, Two-sequence, Two-period, Crossover, Oral Bioequivalence Study of Etodolac Tablets USP 500mg of Ipca Laboratories Limited, India and Etodolac Tablets USP 500mg of Taro Pharmaceutical Industries Ltd., USA in Healthy, Adult, Human Subjects Under Fed Condition.
Brief Title: Bioequivalence Study of Etodolac Tablet USP 500 mg Under Fed Condition
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: IPCA Laboratories Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Ipca/VIN-11/412
Record Dates: First submitted 2012-11-05; First posted 2012-11-28 (Estimated); Last update posted 2012-12-03 (Estimated); Status verified 2012-11

CONDITIONS: Fed
MeSH Terms: conditions — Lecithin Cholesterol Acyltransferase Deficiency | interventions — Etodolac

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Etodolac Tablets USP 500mg (Experimental): Etodolac Tablets USP 500 mg of Ipca Laboratories Limited, India
  Interventions: Drug: Etodolac Tablets USP 500mg
- Etodolac Tablets USP 500 mg (Active Comparator): Etodolac Tablets USP 500 mg of Taro Pharmaceutical Industries Ltd., USA
  Interventions: Drug: Etodolac Tablets USP 500 mg

INTERVENTIONS:
Drug: Etodolac Tablets USP 500mg — 500 mg tablet once a day
  Other Names: Test Product
  Arms: Etodolac Tablets USP 500mg
Drug: Etodolac Tablets USP 500 mg — 500 mg tablet once a day
  Other Names: Reference Product
  Arms: Etodolac Tablets USP 500 mg

SUMMARY:
This is a open Label, balanced, randomized, single dose, two-treatment, two-sequence, two-period, crossover pivotal study. The purpose of this study is to assess the bioequivalence between Test Product and the corresponding Reference Product under fed condition in healthy, adult human subjects.

DETAILED DESCRIPTION:
Objective of this pivotal study was to assess the bioequivalence between Test Product: Etodolac Tablets USP 500 mg of Ipca Laboratories Limited, India and the corresponding Reference Product: Etodolac Tablets USP 500mg of Taro Pharmaceutical Industries Ltd., USA, under fed condition in healthy, adult, human subjects in a randomized crossover study.

The study was conducted with 36 healthy adult subjects. In each study period, a single 500 mg dose of either test or reference was administered to the subjects as per the randomization schedule in each study period with about 240 mL of water at ambient temperature in sitting position.

The duration of the clinical phase was approximately 10 days including washout period of 7 days between administrations of study drug in each study period.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male and non-pregnant female subjects within the age range of 18 to 45 years (both inclusive), at the time of dosing.
2. Subjects' weight within normal range according to normal values for Body Mass Index (18.5 to 24.9 kg/m2) with minimum of 50 kg weight.
3. Subjects with normal health as determined by personal medical and medication history, clinical examination and laboratory examinations within the clinically acceptable reference range.
4. Subjects having normal 12-lead electrocardiogram (ECG).
5. Subjects having normal chest X-Ray (P/A view) whose X-Ray was taken within 6 months prior to the dosing of Period 01.
6. Subjects having negative urine screen for drugs of abuse (including amphetamines, barbiturates, benzodiazepines, marijuana, cocaine, and morphine).
7. Subjects having negative alcohol breath test.
8. Subjects willing to adhere to protocol requirements and to provide written informed consent.
9. Subjects having negative Beta-hCG Pregnancy test (only for female subjects).
10. For Female Subjects:

    * Female of child bearing potential practicing an acceptable method of birth control for the duration of the study as judged by the investigator(s), such as condoms, foams, jellies, diaphragm, intrauterine device (IUD), or abstinence, or
    * Postmenopausal for at least 1 years, or if less than 1 years, then following acceptable contraceptive measures as mentioned above
    * Surgically sterile (bilateral tubal ligation, bilateral oophorectomy, or hysterectomy has been performed on the subject).

Exclusion Criteria:

1. Hypersensitivity to Etodolac or related class of drugs.
2. History or presence of significant cardiovascular, pulmonary, hepatic, renal, gastrointestinal, endocrine, immunological, dermatological, neurological or psychiatric disease or disorder.
3. History or presence of significant alcoholism or drug abuse.
4. History or presence of significant smoking (more than 10 cigarettes or beedi's/day).
5. History or presence of significant asthma, urticaria or other allergic reactions.
6. History or presence of significant gastric and/or duodenal ulceration.
7. History or presence of significant thyroid disease, adrenal dysfunction, organic intracranial lesion such as pituitary tumour.
8. History or presence of cancer.
9. Difficulty with donating blood.
10. Difficulty in swallowing solids like tablets or capsules.
11. Use of any prescribed medication or OTC medical products during last two weeks prior to dosing in period 01.
12. Major illness during 3 months before screening.
13. Participation in a drug research study within past 3 months.
14. Donation of blood in the past 3 months before screening.
15. Consumption of grapefruit juice, xanthine-containing products, tobacco containing products or alcohol within 48 hours prior to dosing.
16. Positive screening test for any one or more: HIV, Hepatitis B and Hepatitis C.
17. History or presence of significant easy bruising or bleeding.
18. History or presence of significant recent trauma.
19. Subjects who have been on an abnormal diet (for whatever reason) during the four weeks preceding the study.
20. Female subjects who are currently on breast feeding.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2012-05; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Cmax | 2 months
  Sampling Hours: Pre-dose and at 0.33, 0.67, 1.00, 1.33, 1.67, 2.00, 2.33, 2.67, 3.00, 4.00, 4.50, 5.00, 6.00, 7.00, 8.00, 10.00, 12.00, 16.00, 24.00 and 36.00 hours post dose.
AUC | 2 months
  Sampling Hours: Pre-dose and at 0.33, 0.67, 1.00, 1.33, 1.67, 2.00, 2.33, 2.67, 3.00, 4.00, 4.50, 5.00, 6.00, 7.00, 8.00, 10.00, 12.00, 16.00, 24.00 and 36.00 hours post dose.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Hardik Dave, M.B.B.S., Principal Investigator — Veeda Clinical Research Pvt. Ltd.
Locations (1):
- Veeda Clinical Research Pvt. Ltd., Ahmedabad, Gujarat, India